CLINICAL TRIAL: NCT04156022
Title: Natural History and Biospecimen Repository for Dystonia; Comprehensive Rating Tools for Cervical Dystonia; Validity & Reliability of Diagnostic Methods & Measures of Spasmodic Dysphonia
Brief Title: Dystonia Coalition Projects
Status: Terminated | Type: Observational
Why Stopped: PI request due to a lack of coordinator availability for study procedures.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: 6301
Record Dates: First submitted 2019-01-08; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Dystonia
Keywords: Cervical dystonia; Cranial dystonia; Limb dystonia
MeSH Terms: conditions — Dystonia; Torticollis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dystonia Coalition is an observational study. — This is not an interventional study.

SUMMARY:
Dystonia is a disorder characterized by excessive involuntary contraction of muscles with repetitive and patterned movements. The primary focal dystonias are the most common type of dystonia and include Limb dystonias (like writer's cramp), Cervical dystonia (spasmodic torticollis), Laryngeal dystonias (like spasmodic dysphonia), and Craniofacial dystonias (like blepharospasm). The purpose of this study is to create resources to help learn more about the primary focal dystonias and to develop and validate various dystonia rating scales.

DETAILED DESCRIPTION:
This collaborative, international effort has two primary goals. The first is to create a biospecimen repository and associated clinical database to be used as a resource for dystonia and related disease research. The second goal is to create and validate various rating scales for focal dystonias to be used during a typical clinical examination. Across sites, the investigators hope to enroll at least 5,000 adult patients.

Subjects of this study will be asked to complete a neurological exam which will be videotaped, complete some questionnaires, and donate a blood sample. A study visit will take between 45 minutes and 1 hour depending upon which portions of the study a subject completes. A subset of subjects will be asked to return no more often than once a year for a one hour follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary dystonia
* To be included in laryngeal dystonia group, nasolaryngoscopy (voice box exam) must have been completed to confirm diagnosis

Exclusion Criteria:

-Any person with secondary dystonia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with dystonia are eligible to participate as long as they are above age 18 and fit the eligibility criteria. The coordinator at the site you contact can tell you more about this.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
To collect clinical data for future studies that will help to understand the varied clinical manifestations, natural history, and pathogenesis of the dystonias. | Through study completion, an average of two years.
  data collected will be demographic and medical information
To create a biospeciman repository as a resource for future research in dystonia and related diseases | Through study completion, an average of two years.
To develop and validate rating scales that can be used to diagnose different forms of dystonia and monitor their severity over time | Through study completion, an average of two years.
  a six phase process will be employed to develop and evaluate a scale that is specifically designed to assess psychiatric co-morbidities in cervical dysplasia (CD)

IPD SHARING:
Plan to Share IPD: Undecided